CLINICAL TRIAL: NCT00420706
Title: A Multi-Dose, Double-Blind, Parallel-Group Study of the Effects of Dose Titration and Administration With Food on the Tolerability of SCA-136 in Healthy Subjects
Brief Title: Study Evaluating SCA-136 Tolerability With Dose Titration and Food
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3153A1-105
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Healthy

INTERVENTIONS:
Drug: SCA-136

SUMMARY:
To evaluate whether the tolerability of SCA-136 is improved by dosing with food or by increasing dose amounts in a step-wise fashion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women, aged 18 to 50 years

Exclusion Criteria:

* Abnormal vital signs, ECG, or lab results

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120
Dates: Start 2006-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of subjects reporting nausea (based on AEs) over the dosing period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Miami, Florida, United States